CLINICAL TRIAL: NCT01912118
Title: Measurement of Nociceptive Index During General Anesthesia in ASA 1-3 Patients Undergoing Elective Surgery Using the Nociception Level (NoL) Index
Brief Title: The Medasense Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medasense Biometrics Ltd (Other)
Responsible Party: Principal Investigator, Albert Dahan, MD, PhD, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NL43511.058.13
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Pain
Keywords: Nociception; General anesthesia
MeSH Terms: conditions — Pain | interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- PROPOFOL ONLY GROUP (Experimental): In this study group measurements will be obtained before intubation or opioid administration. To that end plasma propofol concentration will be increased slowly from 0 to 4 μg/ml in steps of 0.5 μg/mL. After the highest target is reached, the propofol target concentration will be lowered to get a BIS value of 50. After 5-min, the laryngoscope will be inserted into the mouth. Next the laryngoscope will be removed. After 5-min the laryngoscope will be placed again and the patient will be intubated. This will be done without additional administration of muscle relaxant.
  Interventions: Drug: Propofol
- PROPOFOL + REMIFENTANIL TARGET A (Experimental): The subject will be intubated according to the design of group 1. The propofol concentration will be 2-5 μg/kg, aimed at a BIS of 50, with 1 ng/ml remifentanil.
  Interventions: Drug: Propofol; Drug: Remifentanil
- PROPOFOL + REMIFENTANIL TARGET B (Experimental): The subject will be intubated according to the design of group 1. The propofol concentration will be 2-5 μg/kg, aimed at a BIS of 50, with 2 ng/ml remifentanil
  Interventions: Drug: Propofol; Drug: Remifentanil
- PROPOFOL + REMIFENTANIL TARGET C (Experimental): The subject will be intubated according to the design of group 1. The propofol concentration will be 2-5 μg/kg, aimed at a BIS of 50, with 3 ng/ml remifentanil.
  Interventions: Drug: Propofol; Drug: Remifentanil
- PROPOFOL + REMIFENTANIL TARGET D (Experimental): The subject will be intubated according to the design of group 1. The propofol concentration will be 2-5 μg/kg, aimed at a BIS of 50, with 4 ng/ml remifentanil.
  Interventions: Drug: Propofol; Drug: Remifentanil
- PROPOFOL + REMIFENTANIL TARGET E (Experimental): The subject will be intubated according to the design of group 1. The propofol concentration will be 2-5 μg/kg, aimed at a BIS of 50, with 5 ng/ml remifentanil.
  Interventions: Drug: Propofol; Drug: Remifentanil
- PROPOFOL TARGET BIS 30 + REMIFENTANIL TARGET C (Experimental): The subject will be intubated according to the design of group 1. The remifentanil target will be 3 ng/ml remifentanil. The propofol concentration will aim a BIS of 30.
  Interventions: Drug: Propofol; Drug: Remifentanil
- PROPOFOL TARGET BIS 70 + REMIFENTANIL TARGET C (Experimental): The subject will be intubated according to the design of group 1. The remifentanil target will be 3 ng/ml remifentanil. The propofol concentration will aim a BIS 70.
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Propofol — Propofol will be titrated via a target controlled infusion to reach a specific target BIS (as specified in treatment arm)
  Other Names: Diprivan
Drug: Remifentanil — Remifentanil will be provided by a target controlled infusion to a specific effect site concentration (as specified in treatment arm)
  Other Names: Ultiva
  Arms: PROPOFOL + REMIFENTANIL TARGET A; PROPOFOL + REMIFENTANIL TARGET B; PROPOFOL + REMIFENTANIL TARGET C; PROPOFOL + REMIFENTANIL TARGET D; PROPOFOL + REMIFENTANIL TARGET E; PROPOFOL TARGET BIS 30 + REMIFENTANIL TARGET C; PROPOFOL TARGET BIS 70 + REMIFENTANIL TARGET C

SUMMARY:
Despite various efforts there is still the need for adequate monitoring of pain and nociception during anesthesia. In a previous protocol the investigators measured pain responses during anesthesia based on single end-points, eg heart rate,blood pressure and pulse transit time. None of these parameters provided sufficient information regarding nociception. The investigators therefore want to further investigate this matter using a composite parameter, the Nociception Level or NoL. The NoL is a novel index that measures the magnitude of the autonomic response to painful stimuli. The NoL combines information from several physiological parameters, which represent different autonomic pathways. The multi-parameter approach empowered with state-of-the-art signal processing and machine learning techniques. In the current study the investigators will measure the NoL in ASA 1-3 patients undergoing elective surgery under general anesthesia. The investigators will measure NoL responses and the occurrence of patient movement upon the administration of a painful stimulus: Introduction of the laryngoscope, Insertion of the endotracheal tube, Insertion of the gastric tube, Insertion of the bladder catheter and Skin incision.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years;
* Sex: male or female;
* Surgery: Any surgery under general anesthesia;
* ASA status: 1, 2 or 3.

Exclusion Criteria:

* Age: < 18 or > 80 years;
* Unable to give written informed consent;
* Pregnancy/lactation;
* Extreme obesity: BMI > 35;
* Perceived difficult intubation.
* Patients requiring a rapid sequence induction
* Patients on beta-blockers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Nociception level index (NoI) | Between induction and first incision
  The NoL measures the magnitude of the autonomic responses to painful stimuli. The NoL combines information from several physiological parameters which represent different autonomic pathways.

SECONDARY OUTCOMES:
Cardiovascular parameters | Between induction and first incision
  Individual pain related cardiovascular parameters, as heart rate, blood pressure and PPG wave amplitude.
Movement | Between induction and first incision
  Visible occurence of movement during painfull stimuli.
Depth of anesthesia | Between induction and first incision
  Depth of anesthesia is measured by a Bispectral Index monitor. Changes in depth of anesthesia will be recorded during painfull stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD, PhD, Professor, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] Treister R, Kliger M, Zuckerman G, Aryeh IG, Eisenberg E. Differentiating between heat pain intensities: the combined effect of multiple autonomic parameters. Pain. 2012 Sep;153(9):1807-1814. doi: 10.1016/j.pain.2012.04.008. Epub 2012 May 29. PMID 22647429
- [Background] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792